CLINICAL TRIAL: NCT05296057
Title: Pilot Study to Evaluate Virtual Reality Exposure Therapy on People With Epilepsy and Related Anxiety
Brief Title: Pilot to Evaluate VR-Therapy on People With Epilepsy and Related Anxiety
Acronym: AnxEpiVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: York University (Other)
Responsible Party: Principal Investigator, Lora Appel, Post-doc Research Fellow; Assistant Professor, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AnxEpiVR
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Epilepsy; Anxiety Disorders and Symptoms
Keywords: Epilepsy; Anxiety; Virtual Reality; Exposure Therapy; Cognitive Behavioural Therapy (CBT); Neurological Disorder; Psychiatric Disorder; Psychiatric Co-Morbidities; Interictal Anxiety; Mental Health; Panic Disorder; Phobia; Social Phobia; Agoraphobia; Generalized Anxiety; Anticipatory Anxiety; Neurological Diseases; Psychopathology; Non-Pharmacological Intervention; Biomedical Technology; Mental Disorders; Virtual Reality Exposure Therapy
MeSH Terms: conditions — Epilepsy; Anxiety Disorders; Nervous System Diseases; Mental Disorders; Psychological Well-Being; Panic Disorder; Phobic Disorders; Phobia, Social; Agoraphobia; Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: As this is a pilot study, a control will not be included. Findings from this pilot will inform methods for a subsequent larger clinical trial that will include a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants Receiving VR-Exposure Therapy Treatment (Experimental): All participants will be receiving the experimental VR-exposure therapy treatment.
  Interventions: Device: Participants Receiving VR-Exposure Therapy Treatment

INTERVENTIONS:
Device: Participants Receiving VR-Exposure Therapy Treatment — In the baseline interview with an exposure therapy specialist and a member of the research team, participants will be presented with approximately three sets of possible exposure scenarios, each associated with approximately three different scenes that increase in severity level. Through discussion with the exposure therapy specialist, the participant will choose the exposure scenario (out of the three options) that most closely resembles their own epilepsy- or seizure-related fears. As the treatment, the participant will be exposed to the scenes that are associated with their chosen exposure set in a hierarchical manner using an immersive head-mounted display. The participant will work through the three levels of the chosen exposure scenario for approximately two weeks, ideally on each level for four days.

SUMMARY:
Over 28% of people with epilepsy (PwE) struggle from at least one anxiety disorder, making anxiety the most common psychiatric comorbidity in this population. Despite the importance of treating anxiety in PwE, it has not received much research attention and is often unrecognized and untreated. Research has suggested that including exposure therapy (ET) as a part of an anxiety treatment may be helpful for decreasing anxiety in PwE. Research has also shown that Virtual Reality (VR) is an effective and helpful tool for delivering ET in a number of different types of anxiety disorders, such as posttraumatic stress disorder, panic disorder, and social anxiety disorder.

To the investigators' knowledge, no research has been conducted to-date on using VR to deliver ET (VR-ET) in PwE. People with epilepsy have commonly been excluded from VR studies due to the concern that it may trigger seizures in people with photosensitive epilepsy. Although limited research is available on the use of VR in PwE, hesitations regarding the use of VR in this population have not been substantiated and clinicians and researchers are increasingly considering VR for use in this population.

The use of an immersive VR head-mounted display to deliver ET in this population offers several benefits. For example, studies suggest that VR-ET is an especially useful method for customized treatment when it is not safe or practical to do exposures. This is important to consider as it may not be practical to do exposures in-person during times of pandemic, such as the COVID-19 pandemic. Even outside of the pandemic, VR reduces the need for travel, which is difficult for PwE in normal circumstances as driver's licences are typically suspended after a confirmed seizure. Using VR for ET as opposed to traditional ET can also save money and time, and allow for more equitable access to healthcare resources for those who may not live in urban centers.

The investigators designed and will be rigorously evaluating a VR-ET program administered in private residences specific for PwE that focuses on decreasing anxiety that is specifically related to their epilepsy or seizures. This study would be among the first to evaluate VR-ET in this population. This study will also contribute to the limited body of research that currently exists managing comorbid anxiety in PwE as well as the minimal existing literature about fears specifically related to epilepsy or seizures.

The overall primary objective of this study is to report on the feasibility and appropriateness of the protocol and evaluation instruments for use in the subsequent larger clinical trial. The secondary objective is to evaluate whether VR-ET reduces epilepsy- or seizure-related anxiety in PwE. It is hypothesized that PwE will experience decreased levels of epilepsy-related anxiety after undergoing VR-ET. These findings will be used to inform a future randomized controlled trial.

DETAILED DESCRIPTION:
This pilot trial will be a mixed-methods, single-arm study with a target total recruitment of 5 participants. Each participant will take part in: a baseline interview, 12 to 14 days of the intervention, and then a final interview seven days after the last day of the VR-ET.

After obtaining informed consent and before the baseline interview, participants will receive a document that includes a mindfulness strategy, a self-compassion strategy, and a guided imagery technique. Participants will be encouraged to practice these mechanisms before the baseline interview as they will review them with the exposure therapy specialist at that time.

Baseline (T0):

The research coordinator will set up a time convenient to both parties to conduct a semi-structured interview at baseline (T0) with an exposure therapy specialist and a member of the research team over tele- or video-conferencing software. The baseline interview will involve a questionnaire that collects the participant's demographic information as well as information about their history with health and anxiety. In this interview, participants will also verbally respond to the diagnostic protocol for epilepsy-specific anxiety disorders proposed by Hingray et al. (2019).

During the baseline interview, the exposure therapy specialist will also present the participant with three sets of possible exposure scenarios. Each of the three possible sets of exposures will consist of a distinct overarching epilepsy-related fear that is commonly experienced within this population, as determined in previous findings. The same three exposure scenarios will be presented to each participant in their respective baseline interviews and through discussion, the exposure therapy specialist and participant will determine which exposure set fits most aligns with their individual epilepsy-related fears.

As ET is typically delivered in a hierarchical manner, each exposure set will include three levels of scenes. Therefore, after choosing the appropriate exposure set, the exposure therapy specialist and participant will also discuss the most appropriate order in which the three scenes associated with the chosen set should be delivered during the intervention. Participants during the VR-ET intervention will be exposed to the scenes in order of what is least anxiety-provoking for them to most anxiety-provoking. In preparation to run the study, a total of nine 360-degree videos (3 exposure sets x 3 levels) will be included in the AnxiEpi-VR minimal viable product.

After the baseline interview, participants will also provide their baseline scores for two questionnaires over a secure online platform (the Epilepsy Anxiety Survey Instrument (EASI) and the Perceived Stress Scale (PSS)).

The only in-person aspect of T0 will be when a member of the research team visits the participant's residence to set up the VR equipment and teaches them how to use and store the device. In teaching participants how to use the VR head-mounted display (HMD), participants will practice using the device set to a neutral scene that is not expected to provoke anxiety in PwE. After using the VR HMD, participants will complete the VR Induced Symptoms and Effects (VRISE) questionnaire to record their baseline motion sickness tendencies. The VRISE assessment is one of the four domains included in the Virtual Reality Neuroscience Questionnaire (VRNQ) and evaluates the intensity of motion sickness. The three other domains included in the VRNQ (user experience, game mechanics, and in-game assistance) are not relevant to this study and thus, will not be asked. As a lower score on the VRISE assessment suggests greater motion sickness, anyone who scores below 25 on VRISE after using VR with a neutral scene will not be allowed to continue with the study.

Intervention (T1):

The VR-ET intervention will consist of a five-minute exposure session every day for up to 14 days over a one-on-one video-call with a member of the research team. During each session, PwE will be seated in a chair of their choice at their home. Before each exposure, the researcher will remind participants that if they "feel too overwhelmed" during the exposure, they should remove the HMD (therefore ending the exposure, even if they have not performed the exposure for the full 5 minutes yet) and use coping mechanisms that they prepared with the exposure therapy specialist during the baseline interview. Prior to putting on the HMD, the participant will also fill out a Subjective Units of Distress Survey (SUDS) describing their anxiety levels prior to doing the exposure (in other words, their anticipatory anxiety levels). [If a participant's pre-exposure SUDS score is above 70, they will complete an easier exposure instead.] After completing the pre-exposure SUDS, the participant will then put on the HMD and do the exposure for a maximum of five minutes. After performing each exposure for a maximum of five minutes, the participant will immediately repeat the SUDS so that their anxiety in anticipation of performing the exposure can be compared with the anxiety that they feel immediately after performing the exposure. After completing the first post-exposure SUDS, the participant will then complete the Fast Motion Sickness Scale (FMS). The purpose of collecting FMS scores will be to quantitatively measure motion sickness, specifically the general discomfort and nausea components, that participants may have experienced during the VR exposure session. Participants will then provide another SUDS score 10 minutes after completing the exposure so that it can be assessed whether or not their anxiety decreased over time after completing an exposure session (i.e., immediately after the exposure vs 10 minutes after the exposure).

The intent is that each exposure level will be completed everyday for four days, after which the participant will move onto the next level. However, if it is decided based on the predetermined cut-off points of SUDS scores that the participant is not yet ready to move onto the next level, the previous level will be repeated until they are ready. Specifically, the participant must continue to stay at that exposure level until they score 70 or below.

The goal of the study is for participants to habituate to their fears and ultimately experience decreased levels of anxiety. The expectation is that participants' SUDS scores recorded immediately after the exposure will be lower than their SUDS scores recorded prior to starting the exposure. This alone will provide encouragement to participants to continue performing the exposures. It may also decrease unnecessary safety-seeking behaviours. Even if participants' SUDS scores remain high on the first post-exposure SUDS test, the study may still be considered successful if the scores are lower on the 10-minute post-exposure SUDS test and/or participants' follow-up at T2 suggests that they are engaging in less safety-seeking behaviours compared to before they began the VR-ET.

Post-intervention (T2)

One week (seven days) after completing the last exposure session, the participant will have another semi-structured interview with the exposure therapy specialist and/or a member of the research team over tele- or video-conferencing software. The interview will aim at gathering additional feedback about participants' experiences, including their experience with the various devices,the subjective impact of the VR-ET program, and what may be improved about the program. With participants' consent, this interview will be audio-recorded. [Note: the T2 interview is the only aspect of the entire study that may be audio-recorded.]

Over an online secure platform, participants will repeat the EASI and PSS. They will also respond to the Igroup Presence Questionnaire (IPQ), which assesses an individual's subjective experience of being in a virtual environment when they are physically situated in another. Additionally, participants will respond to the System Usability Scale (SUS), which assesses usability of the hardware and software.

The only in-person part of T2 will be when a member of the research team goes to the participant's house to collect the VR equipment.

ELIGIBILITY:
Inclusion criteria:

* Individuals with self-reported epilepsy aged 18-65
* Individuals that identify as having anxiety related to epilepsy
* Individuals that live in the city of Toronto

Exclusion criteria:

* PwE who were ever told by a neurologist that they have photosensitive epilepsy or photoparoxysmal responses
* PwE that ever found, regardless of what a neurologist may have told them, that they have photosensitive epilepsy
* Individuals with open wounds on face
* Individuals with cervical conditions or injuries that would make it unsafe for them to use the VR headset
* Individuals who cannot speak and understand English
* PwE that started an antidepressant or antianxiety drug in the last twelve weeks
* PwE that started using medical marijuana in the last twelve weeks
* PwE that have tonic-clonic seizures more than once a month
* People with psychogenic non-epileptic seizures
* PwE that were ever told by a neurologist that stress might be a seizure trigger for them
* PwE that ever found, regardless of what a neurologist may have told them, that stress may be a seizure trigger for them
* Individuals that have been diagnosed with panic disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Change in baseline scores using the Epilepsy Anxiety Survey Instrument (EASI) | Baseline and post-intervention (i.e., one week after completing the VR-ET intervention)
  The EASI is validated for assessing epilepsy-related anxiety features and severity. The EASI is an 18-item questionnaire and employs a 4-point scale ranging from 0 to 3. Scores range from 0 to 54, where higher scores suggest more severe anxiety.
  Note that by using the EASI, the investigators are simultaneously using the brEASI (brief Epilepsy Anxiety Survey Instrument), which is a validated screening tool for anxiety disorders in PwE. The brEASI is made up of eight items that are already asked in the EASI, also employing a 4-point scale ranging from 0 to 3. Scores range from 0 to 24, where a score greater than or equal to 7 suggests that the participant likely has an anxiety disorder.
Change in baseline scores using the Perceived Stress Scale (PSS) | Baseline and post-intervention (i.e., one week after completing the VR-ET intervention)
  The PSS assesses how one perceives their own stress levels. The PSS is a 14-item questionnaire and employs a 5-point scale with a range of 0 to 4. Scores range from 0 to 56. Higher scores indicate greater perceived stress levels.

SECONDARY OUTCOMES:
Feasibility and appropriateness of the study procedures and evaluation instruments | One week after completing the VR-ET intervention
  Questions during a semi-structured interview at T2 will assess opinions on the device and VR-therapy program experience including: (1) Ease of using the device; (2) Participants' experience with learning how to use the device; (3) Realism of the 360-degree videos; (4) Subjective remarks on whether or not they experience less fear about the scenario that they were exposed to and their avoidance behaviours in relation to that scenario over the past week in the real world; (5) Subjective remarks on how their epilepsy- or seizure- related anxiety in general compares to before they started the VR-exposure therapy program; (5) Aspects of the program that they thought were particularly helpful or unhelpful; and (6) Experience completing the exposure over a video-call with a member of the research team from their home.

OTHER OUTCOMES:
Anxiety levels after each VR-exposure therapy session | Each day of the VR-ET intervention (approximately two weeks)
  Participants will fill out the "Subjective Units of Distress Survey" (SUDS) at the following time points each day in the program that an exposure is completed:
  1. Before the exposure
  2. Immediately after completing the exposure
  3. Ten minutes after completing the exposure
  The SUDS assesses the participant's anxiety levels on a scale of 0-100. The purpose of using the SUDS will be to assess if: the SUDS scores (i.e., levels of anxiety) that are recorded before completing the exposure are lower compared to the SUDS scores that are recorded immediately after completing the exposure; the SUDS scores decrease over the 10-minute post-exposure SUDS; and if participants' overall anxiety progressively decreases over the course of each exposure level.
Changes in safety-seeking behaviours after completing the VR-ET intervention | One week after completing the VR-ET intervention
  The investigators will evaluate if participants' responses in the post-intervention interview suggest that they are engaging in less safety-seeking behaviours after completing VR-ET.

CONTACTS AND LOCATIONS:
Overall Officials: Lora Appel, Ph.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- Home based, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blocher JB, Fujikawa M, Sung C, Jackson DC, Jones JE. Computer-assisted cognitive behavioral therapy for children with epilepsy and anxiety: a pilot study. Epilepsy Behav. 2013 Apr;27(1):70-6. doi: 10.1016/j.yebeh.2012.12.014. Epub 2013 Feb 1. PMID 23376339
- [Background] Deng W, Hu D, Xu S, Liu X, Zhao J, Chen Q, Liu J, Zhang Z, Jiang W, Ma L, Hong X, Cheng S, Liu B, Li X. The efficacy of virtual reality exposure therapy for PTSD symptoms: A systematic review and meta-analysis. J Affect Disord. 2019 Oct 1;257:698-709. doi: 10.1016/j.jad.2019.07.086. Epub 2019 Jul 30. PMID 31382122
- [Background] Hingray C, McGonigal A, Kotwas I, Micoulaud-Franchi JA. The Relationship Between Epilepsy and Anxiety Disorders. Curr Psychiatry Rep. 2019 Apr 29;21(6):40. doi: 10.1007/s11920-019-1029-9. PMID 31037466
- [Background] Maples-Keller JL, Yasinski C, Manjin N, Rothbaum BO. Virtual Reality-Enhanced Extinction of Phobias and Post-Traumatic Stress. Neurotherapeutics. 2017 Jul;14(3):554-563. doi: 10.1007/s13311-017-0534-y. PMID 28512692
- [Background] Munger Clary HM. Anxiety and epilepsy: what neurologists and epileptologists should know. Curr Neurol Neurosci Rep. 2014 May;14(5):445. doi: 10.1007/s11910-014-0445-9. PMID 24652453
- [Background] Newsom-Davis I, Goldstein LH, Fitzpatrick D. Fear of seizures: an investigation and treatment. Seizure. 1998 Apr;7(2):101-6. PMID 9627199
- [Background] Novakova B, Harris PR, Ponnusamy A, Reuber M. The role of stress as a trigger for epileptic seizures: a narrative review of evidence from human and animal studies. Epilepsia. 2013 Nov;54(11):1866-76. doi: 10.1111/epi.12377. Epub 2013 Oct 1. PMID 24117321
- [Background] Siqueira NF, Oliveira FLBB, de Souza EAP. Impaired responsibility dimension of self-esteem of Brazilian adolescents with epilepsy. Epilepsy Behav. 2017 Aug;73:1-5. doi: 10.1016/j.yebeh.2017.05.009. Epub 2017 Jun 9. PMID 28605627
- [Background] Grewe P, Lahr D, Kohsik A, Dyck E, Markowitsch HJ, Bien CG, Botsch M, Piefke M. Real-life memory and spatial navigation in patients with focal epilepsy: ecological validity of a virtual reality supermarket task. Epilepsy Behav. 2014 Feb;31:57-66. doi: 10.1016/j.yebeh.2013.11.014. Epub 2013 Dec 18. PMID 24361763
- [Background] Tychsen L, Thio LL. Concern of Photosensitive Seizures Evoked by 3D Video Displays or Virtual Reality Headsets in Children: Current Perspective. Eye Brain. 2020 Feb 11;12:45-48. doi: 10.2147/EB.S233195. eCollection 2020. PMID 32104130
- [Background] Wang Z, Luo Z, Li S, Luo Z, Wang Z. Anxiety screening tools in people with epilepsy: A systematic review of validated tools. Epilepsy Behav. 2019 Oct;99:106392. doi: 10.1016/j.yebeh.2019.06.035. Epub 2019 Sep 12. PMID 31521915
- [Background] Mula M. Treatment of anxiety disorders in epilepsy: an evidence-based approach. Epilepsia. 2013 Mar;54 Suppl 1:13-8. doi: 10.1111/epi.12101. PMID 23458462
- [Background] Beyenburg S, Mitchell AJ, Schmidt D, Elger CE, Reuber M. Anxiety in patients with epilepsy: systematic review and suggestions for clinical management. Epilepsy Behav. 2005 Sep;7(2):161-71. doi: 10.1016/j.yebeh.2005.05.014. PMID 16054870
- [Background] Gur-Ozmen S, Leibetseder A, Cock HR, Agrawal N, von Oertzen TJ. Screening of anxiety and quality of life in people with epilepsy. Seizure. 2017 Feb;45:107-113. doi: 10.1016/j.seizure.2016.11.026. Epub 2016 Dec 6. PMID 27984808
- [Background] Kotwas I, McGonigal A, Bastien-Toniazzo M, Bartolomei F, Micoulaud-Franchi JA. Stress regulation in drug-resistant epilepsy. Epilepsy Behav. 2017 Jun;71(Pt A):39-50. doi: 10.1016/j.yebeh.2017.01.025. Epub 2017 May 8. PMID 28494323
- [Background] Scott AJ, Sharpe L, Thayer Z, Miller LA, Hunt C, MacCann C, Parratt K, Nikpour A, Wong T, Gandy M. Design and validation of two measures to detect anxiety disorders in epilepsy: The Epilepsy Anxiety Survey Instrument and its brief counterpart. Epilepsia. 2019 Oct;60(10):2068-2077. doi: 10.1111/epi.16348. Epub 2019 Sep 27. PMID 31560136
- [Background] Keshavarz B, Hecht H. Validating an efficient method to quantify motion sickness. Hum Factors. 2011 Aug;53(4):415-26. doi: 10.1177/0018720811403736. PMID 21901938
- [Background] Kourtesis P, Collina S, Doumas LAA, MacPherson SE. Validation of the Virtual Reality Neuroscience Questionnaire: Maximum Duration of Immersive Virtual Reality Sessions Without the Presence of Pertinent Adverse Symptomatology. Front Hum Neurosci. 2019 Nov 26;13:417. doi: 10.3389/fnhum.2019.00417. eCollection 2019. PMID 31849627
- [Derived] Gray HG, Tchao D, Lewis-Fung S, Pardini S, Harris LR, Appel L. Virtual Reality Therapy for People With Epilepsy and Related Anxiety: Protocol for a 3-Phase Pilot Clinical Trial. JMIR Res Protoc. 2023 Jan 24;12:e41523. doi: 10.2196/41523. PMID 36692939
- See also: What is exposure therapy? — https://www.apa.org/ptsd-guideline/patients-and-families/exposure-therapy
- See also: More than seizures: In people with epilepsy, social anxiety affects quality of life — http://www.ilae.org/journals/epigraph/epigraph-vol-21-issue-1-winter-2019/more-than-seizures-in-people-with-epilepsy-social-anxiety-affects-quality-of-life
- See also: Epilepsy and memory — http://practicalneurology.com/articles/2019-oct/epilepsy-memory
- See also: Antidepressant medications — https://www.camh.ca/en/health-info/mental-illness-and-addiction-index/antidepressant-medications
- See also: Igroup Presence Questionnaire (IPQ) — http://www.igroup.org/pq/ipq/index.php